CLINICAL TRIAL: NCT01202942
Title: Smoking Topography and Harm Exposure in a New Potentially Reduced Exposure Product
Brief Title: Use and Harm Exposure in New Low Nicotine Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 805584
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2012-11

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — qing-xin-jie-yu granules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quest (Experimental): Participants smoke Quest cigarettes level 1 for 10 days, followed by level 2 for 10 days, and finally by level 3 for 10 days.
  Interventions: Other: Quest
- Preferred brand (No Intervention): Participants smoke their preferred brand of cigarettes for the duration of the study.

INTERVENTIONS:
Other: Quest — Participants smoke Quest cigarettes level 1 for 10 days, level 2 for 10 days, level 3 for 10 days.
  Arms: Quest

SUMMARY:
The proposed research extends previous research on Quest® cigarette smoking behavior by testing whether compensatory smoking occurs as cigarette nicotine level decreases, and whether, as a result, biomarkers of harm exposure increase. This hypothesis will be tested in 210 smokers who report smoking at least 15 cigarettes per day and have been smoking for at least five years and are not currently interested in quitting, but interested in trying a new cigarette product. Participants will be randomized to one of three conditions: 1) smoke their own preferred brand (control group); 2) smoke Quest® cigarettes in progressively decreasing cigarette nicotine level (step-down); or 3) Quest® cigarette non-step-down condition, where they will smoke Quest® cigarettes in a random order. The study will consist of 4 stages beginning with a 5-day preferred own brand cigarette smoking phase for all participants, followed by one of the three cigarette conditions. For those smoking Quest® cigarettes, cigarette nicotine level will change every 10 days, either in a step-down or random fashion. The primary behavioral outcome is smoking topography, a quantitative measurement of smoke exposure. Alveolar carbon monoxide (CO), a validated assessment of smoke exposure, and urine samples to assess carcinogen exposure, specifically NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol) and 1-HOP (1-hydroxypyrere), and exhaled breath condensate will also be collected at the laboratory visits. At the initiation of the study, participants will view the Quest® print advertisement and complete a survey related to product expectations in order to determine the impact marketing and advertisement has on beliefs, attitudes and behaviors related to Quest® cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Self-report smoking > 15 daily cigarettes.
* Self-report smoking only non-menthol cigarettes.
* Not currently trying to quit smoking, or planning to quit in the next 2 months.
* Interested in trying a new cigarette-like product.

Exclusion Criteria:

* Not meeting any of the inclusion criteria.
* Self-report drinking > 25 alcohol-containing drinks per week.
* Self-report currently using any nicotine replacement products.
* Self-report substance use disorders (abuse or dependence involving alcohol, cocaine, or stimulants, benzodiazepines, not nicotine) in the last 5 years.
* Self-report past history of Axis I psychiatric disorders other than depression
* Self-report myocardial infarct within the past year.
* Females must not be currently pregnant, planning a pregnancy during the study, or currently breastfeeding/lactating.
* Provide a baseline CO reading < 10 ppm

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2007-07; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Smoking topography measures increase as nicotine levels decrease | Every five days over 35 day study participation

SECONDARY OUTCOMES:
Nicotine levels effects on smoking topography | Every 5 days over 35 day study participation.
Whether smokers' inferences from advertising affect smoking behavior | Every 5 days over 35 day study participation.
Whether carbon monoxide boost and biomarkers of harm increase as cigarette nicotine levels decrease | Every 5 days over 35 day study participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tobacco Use Research Center, UPenn, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] DeAtley T, Stone MD, Johnson AC, Mercincavage M, Audrain-McGovern J, Strasser AA. Differences in biobehavioral measures of cigarette smoking by depression symptomology. Addict Behav. 2023 Nov;146:107800. doi: 10.1016/j.addbeh.2023.107800. Epub 2023 Jul 3. PMID 37437421